CLINICAL TRIAL: NCT04010877
Title: Multi-center Phase I/II Clinical Trial of Multiple CAR T Cells for Treating Acute Myeloid Leukemia
Brief Title: Multiple CAR-T Cell Therapy Targeting AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-19004
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; CAR T; CD33, CD123, CLL-1
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple CAR T cells to treat AML (Experimental): Multiple CAR T cells to treat AML
  Interventions: Biological: CLL-1, CD33 and/or CD123-specific CAR gene-engineered T cells

INTERVENTIONS:
Biological: CLL-1, CD33 and/or CD123-specific CAR gene-engineered T cells — Infusion of CLL-1, CD33 and/or CD123-specific CAR-T cells

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of multiple CAR T-cell therapy which combines CAR T cells against CLL-1 with CAR T cells targeting CD123 or CD33 in patients with relapsed and refractory AML. The study also aims to learn more about the function of CAR T cells and their persistency in AML patients.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a malignant disease characterized by the rapid growth of myeloblasts that grow in the bone marrow and interfere with the generation of normal blood cells.

Over the past few years, several groups have demonstrated that CD33 and CD123 CAR T cells can eradicate AML in both preclinical and clinical trials. Nevertheless, relapse after CAR T therapy remains a critical problem in treating AML. Disease relapse can be caused by antigen escape and by the outgrowth of residual leukemia stem cells (LSCs) that are not effectively eliminated by CAR T cells. CLL-1 (C-type lectin-like molecule-1) is a transmembrane glycoprotein, which is overexpressed in LSCs but absent in HSCs (hematopoietic stem cells), suggesting that CLL-1 might be a promising target for novel AML therapy. In this study, we use CLL-1 CAR-T in combination with CD123 and/or CD33 CAR-T as a new strategy to address LSC issue and prevent relapse caused by antigen escape.

The T cells from patients or transplantation donors will be genetically modified with lentiviral CAR vector to recognize specific molecules (CD33, CD123 or CLL-1) expressed on the surface of AML cells. The engineered T cells will be applied to patients through intravenous delivery.

The purpose of this clinical trial is to assess the feasibility, safety and efficacy of multiple CAR-T cell therapy in AML. Another goal of the study is to learn more about the function of CAR T cells and their persistency in the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. Confirmed expression of CLL-1, CD123 and/or CD33 in blast AML by immuno-histochemical staining or flow cytometry.
3. Karnofsky performance status (KPS) score is higher than 80 and life expectancy > 3 months.
4. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: cardiac ejection fraction ≥ 50%, oxygen saturation ≥ 90%, creatinine ≤ 2.5 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, total bilirubin ≤ 2.0mg/dL.
5. Hgb≥80g/L.
6. No cell separation contraindications.
7. Abilities to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
2. Active bacterial, fungal or viral infection not controlled by adequate treatment.
3. Known HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. Pregnant or nursing women may not participate.
5. Use of glucocorticoid for systemic therapy within one week prior to entering the trial.
6. Previous treatment with any gene therapy products.
7. Patients, in the opinion of investigators, may not be able to comply with the study.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion | 1 year
  Treatment-related adverse events are assessed by NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Clinical response | 1 year
  Objective responses (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Ph.D, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China